CLINICAL TRIAL: NCT04237389
Title: Comparative Assessment of Catheter and Thoracoscopic Approaches in Patients With Persistent and Long-standing Persistent Atrial Fibrillation
Brief Title: Thoracoscopic Ablation Versus Catheter Ablation in Patients With Atrial Fibrillation
Acronym: TACAAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center of Surgery, Russia (Other Government)
Responsible Party: Principal Investigator, Revishvili Amiran Shotaevich, M.D., Ph.D., Academician of the Russian Academy of Science, Head of the A.V. Vishnevsky National Medical Research Center of Surgery, National Research Center of Surgery, Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRCSRussia02
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: persistent atrial fibrillation; catheter ablation; thoracoscopic ablation; LAA removal; Box-lesion; ablation index; high-density mapping; hybrid procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation Index guided catheter radiofrequency ablation (Active Comparator): 30 patients, who undergo Ablation Index (AI) guided catheter RF ablation
  Interventions: Procedure: Ablation Index Guided endocardial catheter radiofrequency ablation
- Thoracoscopic surgical epicardial ablation (Active Comparator): 30 patients, who undergo thoracoscopic ablation using "Box-lesion" set
  Interventions: Procedure: minimally invasive thoracoscopic surgical epicardial ablation.

INTERVENTIONS:
Procedure: Ablation Index Guided endocardial catheter radiofrequency ablation — Ablation Index (AI) guided catheter RF ablation with circumferential ablation around the right and left PVs and 2 additional lines between the lower and upper PVs (endoBox-lesion).
  Arms: Ablation Index guided catheter radiofrequency ablation
Procedure: minimally invasive thoracoscopic surgical epicardial ablation. — Description: minimally invasive thoracoscopic surgical epicardial ablation using "Box-lesion" set, which includes isolation of the right and left PVs, roof and posterior wall lines and removal of the LAA.
  Arms: Thoracoscopic surgical epicardial ablation

SUMMARY:
Despite good progress in the management of patients with atrial fibrillation (AF), this arrhythmia remains one of the major causes of stroke, heart failure, sudden death, and cardiovascular morbidity in the world. Furthermore, the number of patients with AF is predicted to rise steply in the coming years.

Even if the amount of antiarrhythmic drugs (AAD) is constantly increasing, there is a group of patients who has AF, resistant to AAD therapy. In such cases they are being offered alternative minimally invasive procedures, such as catheter or thoracoscopic ablation. With the discovery that AF often is initiated and maintained by electrical instability inside and around the pulmonary veins (PV) catheter and thoracoscopic ablation are now widely accepted invasive strategies to cure AF.

Even though the results of both of the procedures are very promising in treating patients with paroxysmal AF, the decision making process, which approach should be used in patients with persistant or LSPAF, is still very controversial.

According to 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS, catheter or surgical ablation should be considered in patients with symptomatic persistent or long-standing persistent (LSP) AF refractory to AAD therapy to improve symptoms, considering patient choice, benefit and risk, supported by an AF Heart Team (IIaC).

Since, there is no actual evidence base, which approach is more effective and save in patients with persistant and LSP AF, the aim of the investigator's study is to evaluate the results of both of the approaches in such group of patients.

DETAILED DESCRIPTION:
The aim of this study is to compare 2 approaches for AF treatment, endocardial catheter isolation of the pulmonary veins (PV) versus minimally invasive thoracoscopic surgical epicardial ablation.

The patients in both groups will be comparable and have persistant or LSP AF only. Patients with previous catheter ablations or any interventions or open heart procedures in the anamnesis will be excluded. The catheter ablation will be Ablation Index-guided, which means that every ablation point will be taken according to ablation quality marker which corporates power, delivery time, contact force (CF), and catheter stability, called Ablation Index (AI). Both of the procedures will be performed by a single identical protocol including wide complete circumferential ablation around the right and left PVs, and additional lines between the lower and upper PVs. The thoracoscopic procedure will be supplemented with removal of left atrial appendage (LAA).

In cases of AF or other atrial tachycardia recurrence after both procedures, every patient will undergo the opposite procedure (for example, if patient after thoracoscopic ablation will be diagnosed an AF recurrence, he will undergo catheter ablation). That is why there will be the third group, the so-called Hybrid procedure group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years old
* Patient has nonparoxismal atrial fibrillation
* Sympthomatic AF
* Patient is refractory to at least one antiarrhythmic drug
* Indications for catheter or thoracoscopic ablation
* Absence of previous failed catheter or surgical AF ablations
* Patients agreement

Exclusion Criteria:

* Patient is younger than 18 years old
* Contraindications for catheter or thoracoscopic ablation
* Any previous heart surgeries (open/interventional)
* Congenital heart diseases
* Paroxismal AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF and other atrial tachycardia | 12 month
  Freedom from AF and other atrial tachycardias, lasting more than 60 sec, determined by 24-hour Holter monitoring.
  Other atrial tachycardias include left atrial flutters, typical atrial flutters
Major adverse cardiac and cerebral events (MACCE) | 12 month
  MACCE include death, stroke, transitory ischemic attack, hemopericarditis, implantation if pacemaker.

SECONDARY OUTCOMES:
Freedom of AAD | 12 month
  Freedom from any AAD and anticoagulation
Postoperative hospitalization duration | 2 month
  The ammount of days after the procedure, wich were spent in the hospital
Decrease in the frequency of AF episodes | 12 month
  Decrease of the ammount of AF episodes

CONTACTS AND LOCATIONS:
Overall Officials: Elena A Artyukhina, Study Chair — A.V. Vishnevsky National Medical Research Center of Surgery
Locations (1):
- A.V. Vishnevsky National Medical Research Center of Surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castella M, Kotecha D, van Laar C, Wintgens L, Castillo Y, Kelder J, Aragon D, Nunez M, Sandoval E, Casellas A, Mont L, van Boven WJ, Boersma LVA, van Putte BP. Thoracoscopic vs. catheter ablation for atrial fibrillation: long-term follow-up of the FAST randomized trial. Europace. 2019 May 1;21(5):746-753. doi: 10.1093/europace/euy325. PMID 30715255